CLINICAL TRIAL: NCT04093466
Title: A Phase 1, Multicenter, Open-label, Dose Escalation/expansion Study Evaluating the Safety, Pharmacokinetics and Preliminary Efficacy of CX1003 (Kanitinib) in the Patients with Relapsed Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of CX1003 (Kanitinib) in Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other); West China Hospital (Other); Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNTN-I-02
Record Dates: First submitted 2019-09-15; First posted 2019-09-18 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CX1003) (Experimental): Treatment will comprise 2 periods: a 4-day single dose period, followed by a period of daily-dose in continuous 28-day treatment cycle (the 1st cycle) or 21-day treatment cycles (the 2nd cycle and beyond).
  Interventions: Drug: CX1003

INTERVENTIONS:
Drug: CX1003 — Oral dose A 4-day single dose period, followed by a period of daily-dose in continuous 28-day treatment cycle (the 1st cycle) or 21-day treatment cycles (the 2nd cycle and beyond) Dosage range: 25 mg, 50mg, 75mg, 100mg,125mg,150mg,175mg
  Other Names: kanitinib

SUMMARY:
CX1003 is a novel multi-target tyrosine kinase inhibitor that is designed to primarily inhibit vascular endothelial growth factor receptor 2 (VEGFR2) and hepatocyte growth factor receptor (HGFR/MET). This study aimed to evaluate the safety, pharmacokinetics, and antitumor activity of CX1003 in patients with refractory advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic solid tumors;
* At least one measurable lesion (spiral CT scan long diameter ≥10 mm or enlarged lymph node short diameter ≥15 mm by RECIST 1.1);
* Documented disease progression after, or refractory to, or intolerant of prior standard or established therapy known to provide clinical benefit for their condition; or documented disease progression within 24 weeks after prior adjuvant/neoadjuvant therapy;
* ECOG PS ≤1;
* Expected overall survival≥12 weeks;

Exclusion Criteria:

* Untreated brain metastases or symptoms of brain metastases cannot be controlled more than 4 weeks;
* Other kinds of malignancies [excluding stage IB or lower grade cervical cancer，noninvasive basal cell or squamous cell cancer, breast cancer with complete remission (CR) > 10 years ,melanoma with CR > 10 years or other malignant tumors with CR > 5 years];
* Hematologic, renal, and hepatic function abnormities as defined below:

Absolute neutrophil count (ANC) <1.5×109 /L or platelet <100×109 /L or hemoglobin <9 g/dL; Total bilirubin > 1.5×the upper limit of normal range(ULN) without liver metastases; total bilirubin > 3×ULN with liver metastases; AST, ALT, ALP >1.5×ULN without liver metastases ; AST, ALT, ALP >5×ULN with liver metastases; Primary hepatocellular carcinoma; Hepatic cirrhosis with Child-Pugh B or C; Serum creatinine >1.5×ULN; History of previous nephrotic syndrome; INR or aPPT >1.5×ULN; Presence of hemorrhage (hemoptysis) , thrombosis，or currently receiving treatment with warfarin, aspirin, low molecular weight heparin (LMWH), or any other anti-platelet drugs (Aspirin ≤100 mg/d for prophylaxis are allowed); •Any of the following gastrointestinal disease: Unable to swallow oral drugs; Need intravenous nutrition; History of a gastric resection; History of treatment for active peptic ulcer disease within 6 months; Clinically significant gastrointestinal bleeding within 3 months; Persistent grade 2 or higher chronic diarrhea despite optimal medical management;

•Any of the following cardiovascular and cerebrovascular disease: Myocardial infarction , severe cardiac arrhythmias, unstable angina, coronary artery disease, congestive heart failure, cerebrovascular accident or TIA within 12 months ; Deep vein thrombosis or pulmonary embolism within 6 months; QTcF >470 msec; Uncontrolled hypertension despite optimal medical management;

* Presence of unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 grade 0 or 1 with the exception of alopecia;
* Involved in other clinical trials within 30 days of enrollment;
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days of enrollment;
* History of organ allograft ;
* Need glucocorticoids or other immunosuppressive agents for immunosuppression (excluding local or inhaled glucocorticoids);
* Uncontrolled ongoing or active infection;
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy;
* Pregnant or lactating women or those who do not take contraceptives, including men;
* Suffering from mental and neurological diseases;
* Any other metabolic dysfunction, abnormal physical examination findings, or clinical laboratory findings;
* Inability to comply with protocol required procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) by NCI CTCAE 5.0: Dose Escalation Stage | First 5 weeks after initial administration of CX1003
  Occurrence of any of the following toxicities was considered DLT if judged by the Investigator to be possibly, probably, or definitely related to the administration of CX1003:
  * Any Grade 3 or higher non-hematologic toxicity (including persisting nausea, vomiting, diarrhea, and electrolyte imbalances despite optimal medical management);
  * Grade 4 neutropenia for >5 consecutive days;
  * Grade 3 or higher febrile neutropenia;
  * Grade 3 or higher neutropenia associated with infection;
  * Grade 4 thrombocytopenia;
  * Grade 3 or higher thrombocytopenia with clinically significant bleeding or that requires a platelet transfusion.
Maximum tolerated dose (MTD): Dose Escalation Stage | First 5 weeks after initial administration of CX1003
  The maximum tolerated dose (MTD) was defined as the highest dose for a given schedule that was expected to cause DLTs in no more than 33% of patients.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile: Cmax | First 5 weeks after initial administration of CX1003
  Parameters: Peak Plasma Concentration (Cmax)
Pharmacokinetics (PK) profile: Tmax | First 5 weeks after initial administration of CX1003
  Parameters: Time to reach the maximum plasma concentration (Tmax)
Pharmacokinetics (PK) profile: T1/2 | First 5 weeks after initial administration of CX1003
  Parameters: Terminal half-life (T1/2)
Pharmacokinetics (PK) profile: AUC | First 5 weeks after initial administration of CX1003
  Parameters: Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics (PK) profile: CL/F | First 5 weeks after initial administration of CX1003
  Parameters: Apparent body clearence from plasma (CL/F)
Pharmacokinetics (PK) profile: Vz/F | First 5 weeks after initial administration of CX1003
  Parameters: Apparent volume of distribution (Vz/F)
Objective Response Rate (ORR) | up to 24 months
  Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.1.
Progression-free survival (PFS) | up to 24 months
  Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.1 or death due to any cause.
Disease Control Rate (DCR) | up to 24 months
  Disease Control Rate (DCR) was defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | up to 24 months
  Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.1.
Safety profile as assessed by the incidence, duration, and severity of adverse events | From first dose of CX1003 to 30 days after last dose
  Incidence, duration, and severity of AEs measured by laboratory assessments and physical findings according to NCI CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No